CLINICAL TRIAL: NCT06554158
Title: A Phase II Study of Post-Resection Radiation Dose and Treatment Site De-Escalation for Favorable Prognosis Human Papilloma Virus (HPV) or p16-Positive Oropharyngeal Cancer
Brief Title: De-escalation of Adjuvant Radiation for Low-Risk HPV Oropharyngeal Cancers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Collaborators: MedStar Georgetown University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00000196
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Oropharynx Cancer
Keywords: HPV; tonsil; base of tongue; soft palate; oropharyngeal cancer
MeSH Terms: conditions — Oropharyngeal Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Radiation dose: 50Gy (Experimental): 50Gy in 25 fractions to the neck at risk for tumor recurrence, excluding the primary site
  Interventions: Radiation: Radiation Therapy

INTERVENTIONS:
Radiation: Radiation Therapy — De-escalation of Adjuvant Radiotherapy

SUMMARY:
The goal of this clinical trial is to learn whether for intermediate-risk patients who have undergone Transoral Robotic Surgery for HPV/p16(+) oropharyngeal cancer and have minimal smoking history, whether these patients can be treated with a lower-than standard dose, with omission of the primary site in the oropharynx. The main questions it aims to answer are:

Does radiotherapy site and dose-de-escalation lead to similar outcomes compared to historical data on tumor control in patients who are treated with standard radiation doses and treatment fields?

Participants will:

Undergo treatment with a lower than standard radiation dose (50Gy in 25 fractions, with either Intensity Modulated Radiation Therapy (IMRT) or proton beam therapy) and to a smaller than standard radiation field (to the neck only, excluding the original site of tumor in the oropharynx)

DETAILED DESCRIPTION:
HPV+ oropharyngeal carcinoma can be treated with either definitive radiotherapy or transoral surgery (TOS, using a predominantly robotic or laser approach), with equivalent oncologic results.23 The proportion of patients who receive definitive radiotherapy or TOS followed by adjuvant radiotherapy (in over 80% of patients) has roughly reached parity. At large academic centers with significant head and neck cancer expertise, the decision to treat with either definitive radiation or TOS followed by adjuvant radiotherapy is driven by non-oncologic considerations most often dictated by anatomic factors such as the presence of a retropharyngeal internal carotid artery, proximity of nodal disease to the carotid artery, involvement of the soft palate, or patient ability to tolerate resection. None of these factors would be expected to affect the probability of oncologic outcomes.

In addition to definitive radiation, the introduction of improved surgical techniques has allowed select patients with oropharyngeal cancer to undergo resection of the primary disease as well as dissection of neck disease as part of their treatment regimen. The utilization of TOS with neck dissection is followed by observation, radiation or chemoradiation based on standard pathologic risk factors such as the presence of perineural invasion, lymphovascular space invasion, close or involved margins, T3-T4 disease, or the presence of multiple involved lymph nodes .24 25 Since over 50% of patients who are treated with TOS are treated with adjuvant radiation utilizing concurrent chemotherapy based on pathologic factors, and over 80% of patients treated with primary TOS are treated with adjuvant radiation of some form, it is important to consider deintensifying treatment for patients with good prognosis cancers.

The most commonly utilized dose in this clinical situation is 60Gy in 30 fractions; however, this is based on literature from smoking-related cancers that suggest that 57.6Gy in 32 fractions would be an acceptable dose for patients with high-risk disease (Peters et al,).

Treatment with adjuvant therapy for TOS patients has involved several deintensification approaches, depending on pathologic factors. Approaches for de-escalation can include decreasing the treatment volume, decreasing radiation dose, or excluding chemotherapy in patients with extracapsular extension.

The Eastern Cooperative Oncology Group ECOG 3311 trial, a phase II randomized study of TOS patients with HPV(+) oropharyngeal cancers is studying dose de-escalation from 60Gy to 50Gy in intermediate-risk patients receiving adjuvant IMRT radiation, but has not yet reported its results. Another approach in the postoperative setting has been using chemotherapy to decrease the dose of radiation used; the Mayo Clinic in Minnesota has reported the use of docetaxel and cisplatin chemotherapy with low-dose radiation (twice daily radiation to 30-36Gy in 20 fractions) without any unexpected recurrences in 80 patients, with locoregional control of 95% and distant control of 94%.

For patients with extracapsular extension (ECE), the addition of concurrent chemotherapy to adjuvant radiation has not shown a benefit in a retrospective series of 152 patients.28 In fact, the aforementioned ECOG 3311 phase II trial of radiotherapy dose de-escalation for adjuvant patients excludes chemotherapy for all these patients, and is de-escalating radiation dose down to 50Gy in this population. A similar approach in patient with ECE ≤1mm is being taken in the SIRS trial from Mt. Sinai with an expected enrollment of 200 patients, which entails de-escalating radiation dose to 50Gy without chemotherapy. The PATHOS trial from the UK will be doing a direct comparison of patients with ECE >1mm, looking at whether chemotherapy can be omitted from this population of higher-risk patients who have predominantly more extensive ECE.

There is no study which we are currently aware that combines the concept of omission of the primary site from the radiation therapy field with dose de-escalation to the nodal bed at risk. A study that combines these concepts found in the literature as well as current clinical trials would therefore be novel and could have a significant of quality-of-life benefit for patients if found to be effective.

A prospective phase II trial at the University of Pennsylvania of 60 patients omitting the primary resection bed while treating the nodal basin with standard doses of adjuvant radiation has demonstrated excellent control rates.33 With 2-year mean follow-up, local control was 98%, regional control 100%, and distant control was 97% Patients were treated to a standard dose of 60-63 Gy. Excluding the primary site led to 1 recurrence in the 60 patients, which was successfully salvaged via surgical resection. There was a 2% gastrostomy dependence rate in this population.

Radiation will involve with a lower than standard radiation dose (50Gy in 25 fractions, with either IMRT or proton beam therapy) and to a smaller than standard radiation field (to the neck only, excluding the original site of tumor in the oropharynx).

ELIGIBILITY:
Inclusion Criteria:

* Patients must be ≥ 18 years of age on the day of signing informed consent.
* Patients must have a diagnosis of p16+ and/or HPV+ squamous cell carcinoma of the oropharynx (including base of tongue, glossotonsilar sulcus, tonsil, soft palate, vallecula, and/or posterior oropharyngeal wall).
* pathologic stage T1-2 N1 M0 (AJCC 8th ed.) stage I or T3 N0-1 M0 stage II (AJCC 8th ed.) SCCA of the oropharynx, with ≤ 5 distinct nodes involved with tumor, ≤ 2mm ECE (extracapsular extension), ≥ 2mm surgical margins at primary site.
* Karnofsky Performance Status (KPS) ≥ 60 within 8 weeks prior to registration.
* neutrophil:lymphocyte ratio ≤ 5 within 8 weeks of registration.
* hemoglobin count ≥ 10 within 8 weeks of registration. The patient may receive transfusion to reach this goal.
* current non-smoker (at least 6 months) with ≤ 15 pack-year smoking history
* start radiation within 8 weeks of resection (6 weeks preferable)
* have undergone resection of the primary site with Transoral Surgery and neck dissection of at least the ipsilateral neck
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
* Ability to understand and willingness to sign a written informed consent.

Exclusion Criteria:

* Perineural invasion at primary site
* Lymphovascular space invasion at primary site
* Level 4 nodal involvement (even if resected)
* Retropharyngeal nodal involvement (even if resected)
* any intact, unresected disease
* nodal disease pathologically invading adjacent neck musculature
* Patients treated via an invasive, non-oral approach to the primary site, including jaw-splitting mandibulotomy with resection or lateral pharyngotomy
* Prior history of malignancy diagnosed within 2 years prior to registration, except for nonmelanomatous skin cancer that has completed treatment and the patient is deemed as being disease-free or Gleason 6 prostate cancer that is undergoing active surveillance.
* Patient with extracapsular extension (ECE) who has not had a biopsy of an ipsilateral neck lymph node that demonstrated squamous cell carcinoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 2 year
  2 year progression free survival, as determined by standard of care physical examination and standard of care surveillance imaging.

SECONDARY OUTCOMES:
Quality of Life (QOL) | 2 year
  Quality of Life will be measured by validated questionnaires relating to Patient Related Outcomes (EORTC QLQ-C30 (version 3). Completed at baseline (at radiotherapy consult), and then approximately at 1-2 weeks, 3 months, 6, 12, 18 and 24 months after completion of RT. A high scale score represents a higher response level.
Local Control Rate | 2 year
  Local Control as determined by standard of care physical examination and standard of care surveillance imaging.
Regional Control Rate | 2 year
  Regional Control as determined by standard of care physical examination and standard of care surveillance imaging
Distant Metastasis-Free Survival (DMFS) | 2 year
  Distant Metastasis-Free Survival as determined by standard of care physical examination and standard of care surveillance imaging.
Overall Survival (OS) | 2 year
  Overall Survival defined as time from start of treatment until end of study or death.
Rate of percutaneous endoscopic gastrostomy (PEG) tube placement | 1 year
  Rate of PEG tube placement and presence of PEG tube at 1 year in patients who are treated with de-escalated adjuvant radiotherapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Medstar Georgetown University Hospital, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: Undecided
all individual data is deidentified